CLINICAL TRIAL: NCT02363127
Title: Subcutaneous Progesterone (Prolutex) Versus Vaginal Progesterone Capsules (Progeffik) for Endometrial Preparation in Fresh Donated Oocytes Recipients: a Randomised, Prospective, Single-blind, Pilot Study
Brief Title: Subcutaneous Progesterone Versus Vaginal Progesterone for Endometrial Preparation in Fresh Donated Oocytes Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Joaquín Llácer, Gynaecologist. Reproductive Medicine Specialist at Instituto Bernabeu, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BER-PRO-2014-01
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-08

CONDITIONS: Infertility
Keywords: Reproductive Techniques; Infertility; Reproductive Techniques Assisted
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolutex (Experimental): Subcutaneous progesterone
  Interventions: Drug: subcutaneous progesterone
- Progeffik (Active Comparator): Vaginal progesterone
  Interventions: Drug: vaginal progesterone

INTERVENTIONS:
Drug: subcutaneous progesterone — subcutaneous progesterone 25 mg/day
  Other Names: Protulex
  Arms: Prolutex
Drug: vaginal progesterone — vaginal progesterone in capsules 200 mg/3 times a day
  Other Names: Progeffik
  Arms: Progeffik

SUMMARY:
Randomised, prospective, investigator-blinded, controlled, single-centre study to assess the impact on the ongoing pregnancy rate with the use of two progesterones with different administration routes, in recipients of fresh embryos from donor oocytes, undergoing endometrial preparation for fresh embryo transfer.

DETAILED DESCRIPTION:
Exploratory study with a control group treated according to our Service's usual therapeutic regimen for the transfer of embryos with donor oocytes.

The controlled ovarian stimulation protocol in oocyte donors is always calculated according to the standard protocol at the Bernabeu Institute. Endometrial preparation will be carried out following the standard protocol of the Bernabeu Institute as follows: the oestrogen will be administered transdermally and patients with maintained ovarian function undergo medical hypophysectomy with depot GnRH agonists administered in the mid-luteal phase of the previous cycle.

On the day of oocyte retrieval, the patient will be randomised: Group A will be administered subcutaneous progesterone 25 mg/day (Prolutex), and Group B will be administered vaginal progesterone in capsules 200 mg/3 times a day (Progeffik).

The embryo transfer will be performed on day 5 of the embryo culture (Day +5). A biochemical pregnancy test beta- hCG and the P4 analysis will be performed 14 days after oocyte retrieval.

All the cycles will be monitored according to the Department's standard criteria, using transvaginal ultrasound to assess embryonic development and endometrial thickness, as well as analytical controls.

The study will be blinded to the investigator. The evaluating professionals will not know if the subject has been administered vaginal progesterone or subcutaneous progesterone. The medication will be delivered by a person who does not participate in the evaluations and who is dedicated to group assignment, to data centralisation, and to delivering the medication.

The aim of this study is to determine if the ongoing pregnancy rate in patients undergoing a fresh embryo transfer cycle with donor oocytes is affected by the progesterone administration route.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged from 18 to 49 years (both inclusive)
* Woman who wishes to become pregnant
* Endometrial thickness greater 7 mm on the day of patient randomisation to one of the progesterone groups
* Six or more donor retrieved oocytes
* Patient programmed for fresh embryo transfer on day +5 of embryo culture
* BMI lower than 30 Kg/m2
* Infertility that justifies treatment with donor oocytes
* Male with no known karyotype alterations
* Semen by ejaculation from either the partner or from a bank
* Uterus able to support embryo implantation and pregnancy
* Absence of pregnancy before starting the embryo transfer cycle
* Has given prior written consent

Exclusion Criteria:

* - Important systemic diseases, endocrine-metabolic abnormalities involving the pituitary, thyroid, adrenals, pancreas, liver or kidney.
* HIV, HBV or HCV seropositivity
* Undiagnosed vaginal bleeding
* Pregnancy, breastfeeding or any contraindication to becoming pregnant
* Malformation of sexual organs incompatible with pregnancy
* Known allergy to progesterone preparations or their excipients
* Current dependence on alcohol, drugs or psychotropic medication
* Concurrent participation in another study
* Concomitant medication that could interfere with the study medication: different hormonal treatments used in the study, except thyroid hormones, antipsychotics, anxiolytics, hypnotics, sedatives, chronic treatment with prostaglandin inhibitors

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate at 12 weeks gestation | 12 weeks
  ongoing pregnancy rate at 12 weeks gestation using subcutaneous progesterone and using vaginal progesterone capsules

SECONDARY OUTCOMES:
progesterone level on the days of the transfer | 5 days
  progesterone level on the days of the transfer
progesterone level on biochemical pregnancy test beta-hCG | 14 days
  progesterone level on biochemical pregnancy test beta-hCG
endometrium thickness on the day of oocyte retrieval | 0 day
  endometrium thickness on the day of oocyte retrieval
endometrium thickness on the day of embryo transfer | 5 days
  endometrium thickness on the day of embryo transfer
endometrium morphology on the day of oocyte retrieval | 0 day
  endometrium morphology (trilaminar pattern and echogenicity) on the day of oocyte retrieval
endometrium morphology on the day of embryo transfer | 5 days
  endometrium morphology (trilaminar pattern and echogenicity) on the day of embryo transfer
implantation rate | 4-5 weeks
  number of embryo sacs at 4-5 weeks (by ultrasound) versus number of embryos transferred
positive biochemical pregnancy test beta- hCG rate | 14 days
  positive biochemical pregnancy test beta- hCG rate at 14 days
clinical pregnancy rate | 4-5 weeks
  rate of patients with embryo any sac with a heartbeat (by ultrasound)
miscarriage rate | 10 weeks
  miscarriage rate in patients with positive biochemical pregnancy test beta- hCG rate on day +14
occurrence of side effects | day 5, day 14, 4-5 days, 10 weeks
  occurrence of side effects associated with progesterone
comfort in relation to the progesterone administration route | 10 weeks
  comfort in relation to the progesterone administration route

OTHER OUTCOMES:
number of uterine contractions per minute | day 5
  number of uterine contractions per minute on the day of embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Joanquin Llacer, Ph, Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Alicante, Spain